CLINICAL TRIAL: NCT03539497
Title: Prognostic Value of Plasma Mitochondrial DNA and Cytochrome C After Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Peter Radsel, Principal investigator, University Medical Centre Ljubljana
Other Study IDs: UKC-KOIIM-c-arrest
Record Dates: First submitted 2018-03-24; First posted 2018-05-29 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest
Keywords: biomarker
MeSH Terms: conditions — Heart Arrest | interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — mitochondrial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biomarker — Plasma mitochondrial DNA, plasma Cytochrome C

SUMMARY:
The aim of the study is to determine prognostic value of plasma mitochondrial DNA and cytochrome C after cardiac arrest.

The study will be conducted in three parts:

1. Determine plasma concentrations of mitochondrial DNA and cytochrome C in healthy population.
2. Determine release profile of mitochondrial DNA and cytochrome C to plasma after cardiac arrest.
3. Determine plasma prognostic value of mitochondrial DNA and cytochrome C after cardiac arrest and compare it with established prognostic methods.

DETAILED DESCRIPTION:
Scientific background

Cardiac arrest is one of leading causes of mortality in developed world. Survival ranges between 15 and 22%. Patients surviving cardiac arrest can have significant neurological impairment. None of currently available diagnostic methods can detect neurological consequences in early post resuscitation period. Biomarkers (NSE - neuron specific enolase, protein S100, GFAP - glial fibrillary acidic protein), imaging (computer tomography, magnetic resonance imaging) and functional studies (EEG - electro encephalography, SSEP - somatosensory evoked potentials) have all shown only limited prognostic value in predicting survival with good neurological outcome after cardiac arrest.

Mitochondrial damage is one of key mechanisms of postresuscitation dysfunction. Elevated values of mitochondrial damage-associated molecular patterns were already linked to worst survival after cardiac arrest and critical illness.

Mitochondrial damage often results in cell death and mitochondrial damage-associated molecular patterns are released into bloodstream. Mitochondrial damage-associated molecular patterns that can be detected in serum or plasma are: mitochondrial DNA, mitochondrial transcription factor A, N-formyl peptides, succinate, cardiolipin, cytochrome C...

With a more sensitive method of early neuroprognostication after cardiac arrest the limited medical resources could be used more effectively in patients with chance of good neurological recovery.

Aim of the study

The aim of this study is to research the role of mitochondrial damage-associated molecular patterns in patients after cardiac arrest.

1. Determine normal plasma values of mitochondrial damage-associated molecular patterns in healthy population.
2. Compare current prognostic procedures of post-resuscitation neurological damage with prognostic value of mitochondrial DNA and cytochrome C in plasma.

Expected results

Due to central role of mitochondria in hypoxic-ischemic tissue damage a greater mitochondrial damage (measured trough release of mitochondrial damage-associated molecular patterns) is expected to have direct correlation with extent of tissue damage (also neurological). Currently published data indicate that patients with higher plasma mitochondrial DNA levels after cardiac arrest have higher mortality. Correlation of mitochondrial damage-associated molecular patterns to extent of neurological damage in survivors of cardiac arrest was not researched yet.

Methods

1. Measurement of measure mitochondrial damage-associated molecular patterns in healthy population (mitochondrial DNA and cytochrome C).
2. Determination of releasing profile of mitochondrial DNA and cytochrome C in survivors of cardiac arrest and establishment of best sample collection time.
3. Calculation of predictive value for survival of cardiac arrest with good neurological outcome for mitochondrial DNA and cytochrome C.

Mitochondrial damage-associated molecular patterns will be measured in samples of plasma. Mitochondrial DNA will be measured using PCR method. Cytochrome C will be measured using ELISA.

ELIGIBILITY:
Inclusion Criteria:

* unconscious after cardiac arrest
* therapeutic hypothermia

Exclusion Criteria:

* expected survival less than 24h

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Unconscious patients after cardiac arrest treated with therapeutic hypothermia.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of plasma mitochondrial DNA and cytochrome C with survival with good neurological outcome (CPC 1 and 2) at hospital discharge | In hospital mortality, 30days
  Relationship between plasma mitochondrial DNA and cytochrome C with neurological damage after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Marko Noč, MD, Study Chair — UMC Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greer DM, Rosenthal ES, Wu O. Neuroprognostication of hypoxic-ischaemic coma in the therapeutic hypothermia era. Nat Rev Neurol. 2014 Apr;10(4):190-203. doi: 10.1038/nrneurol.2014.36. Epub 2014 Mar 11. PMID 24614515
- [Background] Girotra S, Chan PS, Bradley SM. Post-resuscitation care following out-of-hospital and in-hospital cardiac arrest. Heart. 2015 Dec;101(24):1943-9. doi: 10.1136/heartjnl-2015-307450. Epub 2015 Sep 18. PMID 26385451
- [Background] Arnalich F, Codoceo R, Lopez-Collazo E, Montiel C. Circulating cell-free mitochondrial DNA: a better early prognostic marker in patients with out-of-hospital cardiac arrest. Resuscitation. 2012 Jul;83(7):e162-3. doi: 10.1016/j.resuscitation.2012.03.032. Epub 2012 Apr 7. No abstract available. PMID 22490673
- [Background] Rodrigues Filho EM, Ikuta N, Simon D, Regner AP. Prognostic value of circulating DNA levels in critically ill and trauma patients. Rev Bras Ter Intensiva. 2014 Jul-Sep;26(3):305-12. doi: 10.5935/0103-507x.20140043. PMID 25295826
- [Background] Nakahira K, Hisata S, Choi AM. The Roles of Mitochondrial Damage-Associated Molecular Patterns in Diseases. Antioxid Redox Signal. 2015 Dec 10;23(17):1329-50. doi: 10.1089/ars.2015.6407. Epub 2015 Aug 17. PMID 26067258